CLINICAL TRIAL: NCT03384563
Title: Effect of Dexmedetomidine on the Minimum Alveolar Concentration of Sevoflurane
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Rahul Baijal, Associate Professor, Baylor College of Medicine
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: H-37186
Record Dates: First submitted 2017-12-19; First posted 2017-12-27 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Pediatric Anesthesia
Keywords: pediatric; anesthesia; dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (9):
- Dexmedetomidine 0.5 mcg/kg 1-6 months (Active Comparator): Precedex 0.5mcg/kg intravenous administered over 10 minutes prior to surgical procedure. Assigned sevoflurane concentration.
  Interventions: Drug: Dexmedetomidine
- Dexmedetomidine 1 mcg/kg 1-6 months (Active Comparator): Precedex 1 mcg/kg intravenous administered over 10 minutes prior to surgical procedure. Assigned sevoflurane concentration.
  Interventions: Drug: Dexmedetomidine
- Dexmedetomidine 0.5 mcg/kg 6-12 months (Active Comparator): Precedex 0.5mcg/kg intravenous administered over 10 minutes prior to surgical procedure. Assigned sevoflurane concentration.
  Interventions: Drug: Dexmedetomidine
- Dexmedetomidine 1 mcg/kg 6-12 months (Active Comparator): Precedex 1 mcg/kg intravenous administered over 10 minutes prior to surgical procedure. Assigned sevoflurane concentration.
  Interventions: Drug: Dexmedetomidine
- Placebo 6-12 months (Placebo Comparator): Saline intravenous administered over 10 minutes prior to surgical procedure. Assigned sevoflurane concentration.
  Interventions: Drug: Dexmedetomidine
- Dexmedetomidine 0.5 mcg/kg 1-3 years (Active Comparator): Precedex 0.5mcg/kg intravenous administered over 10 minutes prior to surgical procedure. Assigned sevoflurane concentration.
  Interventions: Drug: Dexmedetomidine
- Dexmedetomidine 1 mcg/kg 1-3 years (Active Comparator): Precedex 1 mcg/kg intravenous administered over 10 minutes prior to surgical procedure. Assigned sevoflurane concentration.
  Interventions: Drug: Dexmedetomidine
- Placebo 1-3 years (Placebo Comparator): Saline intravenous administered over 10 minutes prior to surgical procedure. Assigned sevoflurane concentration.
  Interventions: Drug: Dexmedetomidine
- Placebo 1-6 months (Placebo Comparator): Saline intravenous administered over 10 minutes prior to surgical procedure. Assigned sevoflurane concentration.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine 9 arms
  Other Names: Precedex

SUMMARY:
The purpose of this protocol is to determine the effect of two clinically applicable Dexmedetomidine dosages (0.5mcg/kg and 1mcg/kg) on the minimum alveolar concentration (MAC) of Sevoflurane in children between the age ranges of: 1-6 months; 6-12 months of age and 12 months-36 months years of age.

DETAILED DESCRIPTION:
The anesthetic potency of an inhalational anesthetic is measured by the minimum alveolar concentration (MAC), or the dose required to suppress movement to a surgical stimulus in 50% of patients. This measure of potency may also be used to assess the effects of other agents on the MAC of the inhalational agent. Sedative agents reduce MAC of inhalational anesthetic agents. Two human adult studies have shown that Dexmetomidine decreased the minimum alveolar concentration of Isoflurane and Sevoflurane. Age has an important effect on the MAC of inhalational anesthetics in children. Sevoflurane is a commonly used polyflourinated methyl ether with a low blood:gas partition coefficient, which facilitates a rapid increase in alveolar and tissue anesthetic partial pressures and subsequent rapid emergence from anesthesia. Additionally, Sevoflurane is non-stimulating to airway reflexes facilitating smooth inhalational induction of anesthesia. The MAC of Sevoflurane is also dependent on age with the MAC in neonates (<28 days) 3.3%, infants between 6-12 months of age 3.2%, and infants 6-12 months of age and children 1-12 years of age 2.5%. MAC is affected by several factors. Hypothermia, hyponatremia, hypo-osmolality, metabolic acidosis, hypoxia, hypercarbia, anemia, pregnancy, nitrous oxide, opioids, propofol, benzodiazepines, and acute alcohol use decrease MAC whereas hyperthermia, cocaine, amphetamines, hypernatremia, chronic alcohol use increase MAC. Dexmetomidine is an alpha-2 agonist that has been used as a premedication, an adjunct to analgesia, and an adjunct to general inhalational anesthesia. Alpha-2 adrenergic agonist additionally decease the stress response to surgery. Alpha-2 adrenergic agonists have sedative, hypnotic, and analgesic properties and have been reported to decrease the amount of other sedative, analgesic, and general inhalational anesthetics in not only animal studies but also human studies. A concentration-response relationship has been reported in adults receiving Dexmedetomidine using the visual analog scale (VAS) sedation scale (0-100) with a 0 as very alert and 100 as very sedated. A score of 40 correlated with a Dexmedetomidine concentration of 0.7mcg/mL and a score of 60 with a plasma concentration of 1.2mcg/mL. The sedated target concentration from a pooled population of children and neonates has been reported to be between 0.4 and 0.8 mcg/mL. Additionally, a plasma concentration of 0.6mcg/mL has been estimated as satisfactory for sedation in the adult ICU. Inhalational anesthetics have been shown to cause neuroapoptosis and neurodegenerative changes in various animal models; however, the human data from retrospective and epidemiologic studies in children exposed to inhalational anesthetics is inconclusive. There are ongoing trials to determine the effect of exposure from inhalational anesthetics on neurodevelopment outcomes. There is emerging evidence that Dexmedetomidine is not associated with neuroapoptosis or other neurodegenerative changes. Dexmedetomidine has actually been shown to attenuate Isoflurane-induced neurocognitive impairment in neonatal rats. There is no information regarding the reduction of MAC of Sevoflurane in children with clinically applicable Dexmetomidine dosing regimens. Additionally, determining the degree of reduction of Sevoflurane MAC by Dexmedetomidine may be helpful in providing an alternative anesthetic regimen such as the routine use of Dexmedetomidine and Sevoflurane in order to decrease the potential neuroapoptotic effects of inhalational anesthetic agents.

ELIGIBILITY:
Exclusion Criteria:

1. Interstitial lung disease, chest wall disease, or bronchospastic disease with no flare-ups in the past 2 weeks of presentation
2. History of difficult intubation or ventilation
3. Airway malformation
4. Congenital heart disease
5. Cardiac arrhythmias
6. Central nervous system disease, including developmental delay, cerebral palsy, or seizure disorder
7. History of or family history of malignant hyperthermia
8. Electrolyte disorders
9. Gastrointestinal disease
10. Hepatic dysfunction
11. Renal dysfunction
12. Metabolic disease, such as diabetes
13. Obesity, defined as a body mass index greater than the 95% percentile for age
14. Preterm infant (less than 37 weeks gestational age) 15. Use of any medications (anticonvulsants, opioids, benzodiazepines, antibiotics, antihistamines drugs that induce hepatic enzymes) that may affect MAC.

Inclusion Criteria

All patients age 1 month- 3 years presenting for surgery.

Ages: 1 Month to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2018-02-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Movement | Immediately following skin incision
  The study is completed after assessment of patient movement with skin incision

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Baijal, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No